CLINICAL TRIAL: NCT01667809
Title: Cognitive Behavior Therapy Versus a Return to Work Intervention for Sick-listed Patients With Subclinical Common Mental Illness in Primary Care: a Randomized Controlled Trial
Brief Title: CBT vs RTW Intervention for Patients With Common Subclinical Mental Illness in Primary Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Erik Hedman, Principal investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GVC CBT vs RTW II
Record Dates: First submitted 2012-08-10; First posted 2012-08-17 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Anxiety Disorders; Major Depression; Stress Disorders; Primary Insomnia
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder, Major; Stress Disorders, Traumatic; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy; Return to Work

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavior Therapy (Active Comparator): As the trial will include several different common subclinical mental disorders, the cognitive behavior therapy used in the study will be based on the protocols with best empirical support. Cognitive behavior therapy entails psychoeducational components, i.e. the patient is learns about the disorder and how to view it from a cognitive behavioral perspective. The most important part of the treatment is systematic behavior changes often targeted at exposure to feared stimuli. This is combined with cognitive interventions targeted at challenging negative automatic thoughts. All treatments will be delivered by licensed psychologists.
  Interventions: Behavioral: Cognitive behavior therapy
- Return to work (Experimental): Participants randomized to this arm will receive an experimental treatment, based in cognitive behavioral therapy, with primary aim to help patients return to work. Interventions are aimed at solving work-related problems and comprises problem-solving training and systematic employer-patient meetings aimed at facilitating a gradual return to the workplace. Licensed psychologists deliver all treatments.
  Interventions: Behavioral: Return to work

INTERVENTIONS:
Behavioral: Cognitive behavior therapy — Cognitive behavior therapy entails psychoeducational components, i.e. the patient is learns about the disorder and how to view it from a cognitive behavioral perspective. The most important part of the treatment is systematic behavior changes often targeted at exposure to feared stimuli. This is combined with cognitive interventions targeted at challenging negative automatic thoughts. All treatments will be delivered by licensed psychologists.
  Arms: Cognitive Behavior Therapy
Behavioral: Return to work — Participants randomized to this arm will receive an experimental treatment, based in cognitive behavioral therapy, with primary aim to help patients return to work. Interventions are aimed at solving work-related problems and comprises problem-solving training and systematic employer-patient meetings aimed at facilitating a gradual return to the workplace. Licensed psychologists deliver all treatments.
  Arms: Return to work

SUMMARY:
Background: Common mental illness, such as anxiety disorders and depression, is the main cause for sick leave in Sweden. Cognitive behavior therapy (CBT) has been shown to be effective in alleviating target symptoms of these disorders, but its effect on sick leave rates has not been sufficiently addressed. The investigators have developed an intervention called return to work (RTW), which is based in cognitive behavioral theory, that has a primary aim of helping sick-listed patients with common mental illness return to work. This new treatment has not been evaluated in a randomized controlled trial.

Aims: The aim of this study is to investigate the effect of CBT and RTW for subclinical common mental illness in a randomized controlled trial conducted in primary care. Participants will be randomized to diagnosis specific CBT (n=50), RTW (n=50. Main outcomes are days of sick leave and clinician severity rating of psychiatric symptoms. This study could contribute to new knowledge regarding how to best treat patients on sick leave with mild common mental illness.

ELIGIBILITY:
Inclusion Criteria:

* Have been on sick leave (at least 50%) for at least 1 month and not more than 6 months
* Have subclinical levels of anxiety disorder diagnosis (obsessive compulsive disorder, social phobia, panic disorder, generalized anxiety disorder, post-traumatic stress disorder, specific phobia), or/and major depression, or/and maladaptive stress reaction, or/and primary insomnia. Severity measured by clinical severity rating (CSR) 2-3 for mild subclinical level

Exclusion Criteria:

* A higer score than 3 on the Clinician severity rating scale
* A lower score than 2 on the Clinician severity rating scale

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Sick leave | 1 year
  Number of days on sick leave
Clinician Severity Rating (CSR) | Baseine, post-treatment (12 weeks on average), 26 week follow-up, 52 week follow-up
  Change in CSR at post-treatment, 26 week follow-up, and 52 week follow-up compared to baseline.

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale-Self-report (MADRS-S) | Baseline, post-treatment (12 weeks on average), 26 week follow-up, 52 week follow-up
  Change in MADRS-S at post-treatment, 26 week follow-up, and 52 week follow-up
Insomnia Severity Index (ISI) | Baseline, post-treatment (12 weeks on average) 26 week follow-up, 52 week follow-up
  Change in ISI at post-treatment, 26 week follow-up, and 52 week follow-up
Health Anxiety Inventory (HAI) | Baseline, post-treatment (12 weeks on average), 26 week follow-up, 52 week follow-up
  Change in HAI at post-treatment, 26 week follow-up, and 52 week follow-up
Perceived Stress Scale (PSS) | Baseline, post-treatment (12 weeks on average), 26 week follow-up, 52 week follow-up
  Change in PSS at post-treatment, 26 week follow-up, and 52 week follow-up
Trimbos and Institute of Technology Cost Questionnaire for Psychiatry (TIC-P) | Baseline, post-treatment (12 weeks on average), 26 week follow-up, 52 week follow-up
  Change in TIC-P at post-treatment, 26 week follow-up, and 52 week follow-up
Quality of Life Inventory (QOLI) | Baseline, post-treatment (12 weeks on average) 26 week follow-up, 52 week follow-up
  Change in QOLI at post-treatment, 26 week follow-up, and 52 week follow-up
EuroQol-5 dimension (EQ5D) | Baseline, post-treatment (12 weeks on average) 26 feel follow-up, 52 week follow-up
  Change in EQ5D at post-treatment, 26 week follow-up, and 52 week follow-up
Sheehan Disability Scales (SDS) | Baseline, post-treatment (12 weeks on average), 26 week follow-up, 52 week follow-up
  Change in SDS at post-treatment, 26 week follow-up, and 52 week follow-up
Self-rated health 5 (SRH-5) | Baseline, post-treatment (12 weeks on average), 26 week follow-up, 52 week follow-up
  Change in SRH-5 at post-treatment, 26 week follow-up and 52 week follow-up
Obsessive Compulsive Inventory-Revised (OCI-R) | Baseline, post-treatment (12 weeks on average), 26 week follow-up, 52 week follow-up
  Change in OCI-R at post-treatment, 26 week follow-up, and 52 week follow-up. Disorder specific.
Liebowitz Social Anxiety Scale Self-report (LSAS-SR) | Baseline, post-treatment (12 weeks on average), 26 week follow-up, 52 week follow-up
  Change in LSAS-SR at post-treatment, 26 week follow-up, and 52 week follow-up. Disorder specific.
Panic Disorder Severity Scale Self-rated (PDSS-SR) | Baseline, post-treatment (12 weeks on average), 26 week follow-up, 52 week follow-up
  Change in PDSS-SR at post-treatment, 26 week follow-up, and 52 week follow-up. Disorder specific.
Penn-State Worry Questionnaire (PSWQ) | Baseline, post-treatment (12 weeks on average), 26 week follow-up, 52 week follow-up
  Change in PSWQ at post-treatment, 26 week follow-up, and 52 week follow-up. Disorder specific.
Post Traumatic Stress Disorder Symptom Scale-Self report (PTSDSS) | Baseline, post-treatment (12 weeks on average), 26 week follow-up, 52 week follow-up
  Change in PTSDSS at post-treatment, 26 week follow-up, and 52 week follow-up. Disorder specific.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet and Gustavsberg primary care center, Stockholm, Stockholm County, Sweden